CLINICAL TRIAL: NCT03201588
Title: A Randomized Intervention, Multi-Center Study to Determine the Role of Fatty Acids in Serum in Preventing Retinopathy of Prematurity (MDM)
Brief Title: Multi-Center Study to Determine the Role of Fatty Acids in Serum in Preventing Retinopathy of Prematurity (MDM)
Acronym: MDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 303-11
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Ophthalmological Disorder
Keywords: Retinopathy of Prematurity
MeSH Terms: conditions — Eye Diseases; Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: A randomized intervention study of 105+105 (number based on power analysis regarding up to date ROP frequency, see 5.1 and 11.1) infants without major malformations born with a gestational age less than 28 weeks + 0 days will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulaid (Experimental): Formulaid 2:1 Arachidonic acid/Docosahexaenoic acid (AA/DHA). Enteral supplement of AA (0,1-1ml) (100mg(kg/day) and DHA (50mg/kg/day) from birth to 40 weeks postmenstrual age in addition to conventional parenteral fatty acid treatment with Clinoleic
  Interventions: Dietary Supplement: Formulaid
- Clinoleic (No Intervention): Sterile fat emulsion [containing a mixture of refined olive oil (approximately 80%) and refined soya oil (approximately 20%)] 200 g, egg lecithin (purified egg phospholipids) 12 g, glycerol 22.5 g, sodium oleate 0.3 g and Water for Injections to 1,000 mL (final pH between 6.0-8.0).
  One of the active ingredients, soya oil, contains ascorbyl palmitate as an antioxidant (free radical scavenger), in the concentration of 0.15 mg/g of oil.

INTERVENTIONS:
Dietary Supplement: Formulaid — Arachidonic acids (AA) Docosahexaenoic Acids(DHA) 2:1
  Arms: Formulaid

SUMMARY:
The study is a Randomized Intervention, Multi-Center Study to Determine the Role of Fatty Acids in Serum and Breast Milk in preventing Retinopathy of Prematurity Subjects who meet all inclusion and none of the exclusion criteria will be enrolled into the study. Upon entry into the study, subjects will be randomized and given a unique subject number.

A randomized intervention study of 105+105 (number based on power analysis regarding up to date ROP frequency, see 5.1 and 11.1) infants without major malformations born with a gestational age less than 28 weeks + 0 days will be performed.

DETAILED DESCRIPTION:
Every year around 10-12 % of all infants in Europe and the USA are born prematurely which results in 950000 preterm infants per year (500000 in Europe and 450000 in USA). Direct complications of preterm birth account for one million deaths each year worldwide, and preterm birth is a risk factor in over 50% of all neonatal deaths. In addition, preterm birth can result in a range of long-term complications in survivors, with the frequency and severity of adverse outcomes rising with decreasing gestational age and decreasing quality of care. The annual costs, beside patient suffering and parental emotional stress, of preterm care in USA amounts to 26,2 billion United States dollar in terms of immediate neonatal intensive care, subsequent long-term complex health care needs, as well as lost economic productivity.

Possible problems that may occur after a preterm birth are:

Organ disorders (intestine, heart, lung - BPD and asthma), ears (hearing problems), eyes (ROP and visual problems).

Feeding problems and failure to thrive, Poor general growth,Physical disabilities such as cerebral palsy,Cognitive impairment,Learning disability or behavioral problems such as attention deficit (ADD) or autism spectrum disorders. Of infants born extremely prematurely, i.e. at less than 28 weeks gestation or with extremely low birth weight (<1000 g), 20 - 30% may show developmental disorders requiring treatment (3, 4). Impaired cognitive development and abnormal behavior may cause problems at school; in some countries the percentage of learning difficulties in the preterm population is as high as 25%.

Much has been done to improve neonatal care e.g. target levels for oxygen saturation has been an issue for extensive discussions and clinical trials. In fact, the optimal oxygen saturation level for preterm infants has been called "a moving target", fluctuating almost as much as our patients oxygen saturation levels. Reaching a consensus on what these levels should be is still a work in progress. Nutrient delivery is another important and central area of neonatal care which is closely associated with morbidity outcome, and is in need of evidence-based guidelines. The project therefore aims to improve nutrient delivery to prevent or reduce the development of preterm disabilities.

There is a long tradition in neonatology to develop national and in some cases local guidelines for care in each individual Neonatal Intensive Care Unit (NICU). This has resulted in a wide range of treatment approaches and experience-based strategies. These approaches may differ between countries and hospitals and even between neonatologists at the same hospital. There is, for example, a fragmented approach and incomplete compliance to guidelines for nutrient delivery, one important medical parameter tightly associated with neonatal morbidities. Although over 3000 randomized controlled trials have been reported in the field of neonatology, few interventions have yet been subjected to unbiased evaluation.

Available nutritional fatty acid guidelines are not evidence-based and neither optimal composition nor amounts needed to meet the demands of these immature infants are known. What is known is that most infants born extremely preterm develop a large energy deficit resulting in poor neonatal growth. Many experience moderate hyperglycemia associated with lipid infusion. Hyperglycemia is a strong risk factor for preterm mortality as well as for ROP and other disorders of prematurity. With commonly used lipid solutions, preterm new-borns experience a rapid decline in blood fatty acid proportions of the long chain polyunsaturated fatty acids (LCPUFA), Arachidonic acid (AA) and DHA, as compared to the intra-uterine situation.

In Sweden, approximately 300 infants are born extremely preterm i.e. before 28 gestational weeks yearly. With modern neonatal care, infants born as early as at 23-24 weeks of gestation, in the second trimester of gestation, have more than 50% chance of survival. The third trimester is a period of intense growth and differentiation of the central nervous system (CNS) of which the retina is a part, with rapid formation of synapses and dendritic spines and development of retinal photoreceptor cells. During this fetal time period AA and DHA are selectively transferred from the mother to her fetus and blood fractions of DHA increase above maternal values. AA fractions are high, twice those of the mother, from at least 24 weeks of gestation. After very preterm birth, the fractions of AA and DHA fall. In utero glucose, not lipid is the main source of energy and the LCPUFAs transferred during the third trimester play important structural and functional roles in membranes of the central nervous system and most other organs.

DHA, which is an omega-3 LCPUFA is derived from algae and oily fish is the pre-dominant fatty acid of membrane phospholipids in the brain grey matter and the retina, especially its rod outer segments. DHA is not merely a structural component of cell membranes but essential for proper function of membranes. Since the capacity to synthesize DHA is limited in humans and especially in infants, it needs to be provided in the diet. Dietary DHA is needed for optimal functional maturation of the retina and visual cortex, it is a major component at the synaptic site, modulating the uptake and release of neurotransmitters. Absolute accretion of DHA in the brain is greater before than after term and DHA is also accumulated in adipose tissue. In addition, omega-3 LCPUFA has the potential to reduce oxidative stress, deranged glucose metabolism and inflammation.

While many studies have focused on DHA and its role in fetal and neonatal development, few studies have addressed the role of the omega-6 LCPUFA AA during fetal life and after preterm birth. Like DHA, AA is an important component of cell membranes. Altered cell membrane composition results in altered cell function. AA is abundant in the vascular endothelium and in glia where it plays different roles than DHA which is especially abundant in retinal rod outer segments and in synapses and brain grey matter. In the retina AA metabolites contribute to neurovascular coupling i.e. modulation of blood flow with neuronal activity. Metabolites of AA both stimulate and inhibit inflammation and angiogenesis. In addition, AA is involved in blood vessel tonus control with AA derivatives mediating both vessel relaxation and contraction. Low AA concentrations are associated with late onset sepsis in preterm infants. Improved development of very preterm infants fed twice as much AA as DHA than of infants fed equal amounts of AA and DHA was recently reported.

After extremely preterm birth energy expenditures increase, oral intake often takes some weeks to establish and total parenteral nutrition (TPN) is invariably required during the initial postnatal weeks. After birth lipids are the main source of energy, initially as integral part of administered TPN.

Preterm infants treated with soy and olive oil based parenteral lipid solutions (Intralipid and Clinoleic) have low levels of LCPUFAs and increased supply of DHA has been recommended. It has been demonstrated that low DHA levels are associated with compromised fetal insulin sensitivity and insulin resistance in preterm infants is common and strongly associated with neonatal morbidity. Few studies have examined associations between low AA and preterm neonatal morbidities.

One of the most severe morbidities affecting preterm infants is sight threatening ROP, a disorder characterized by reduced retinal vascularization followed by pathologic neovascularization which can lead to retinal detachment and blindness similar to diabetic retinopathy. ROP develops during the neonatal period and outcome is available around term age (40 postmenstrual weeks), which makes it a useful marker for short term outcome of neurovascular development in interventional studies.

In animal studies, a diet rich in omega-3 LCPUFAs reduced pathologic retinal neovascularization in oxygen induced retinopathy, through reduction of inflammatory mediators and attenuation of endothelial cell activation.

In two recent studies, the frequencies of ROP needing treatment as well as cholestasis were significantly reduced when a solution containing fish oil (SMOFlipid) was provided compared to Clinoleic in preterm infants with birth weight 1250 grams. In addition, ROP frequency was reduced in infants receiving SMOFlipid as compared to those receiving Intralipid. No randomized controlled trial comparing convention-al fatty acid administration without and with supplementation of AA and DHA from birth with regard to ROP has been published.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be permitted into this study:

* Signed informed consent from parents/guardians;
* Subject must be born before 28 weeks of gestation

Exclusion Criteria:

Subjects presenting with any of the following will be excluded from the study:

* Detectable clinical gross malformation;
* Known or suspected chromosomal abnormality, genetic disorder, or syndrome, according to the investigator's opinion;
* Clinically significant neuropathy, nephropathy, retinopathy, or other micro or macrovascular disease requiring treatment, according to the investigator's opinion
* Any other condition or therapy that, in the investigator's opinion, may pose a risk to the subject or interfere with the subject's ability to be compliant with this protocol or interfere with interpretation of results.

Ages: 22 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Investigate whether enteral administration of AA and DHA in addition to commonly used regimes with parenteral olive based lipid emulsion (Clinoleic) compared to Clinoleic alone prevents the sight threatening disease Retinopathy of Prematurity (ROP). | When the retina is fully vascularised, i.e approximately 40 postmenstrual weeks.
  Fatty Acids content (AA/DHA) in children with Retinopathy of Prematurity, change from baseline to 40 weeks postmenstrual weeks. Analyses of phospholipids witch can be done on small amount of blood, is relatively intensitive to short term fluctuations in intake and mirror the composition of many membranes in the body. The analyses will be made by using gas-liquid-chromatography. The method has a coefficient of variability of 1-3% for the Fatty Acids concerned.

SECONDARY OUTCOMES:
Postnatal serum fatty acid composition in preterm infants with and without AA:DHA supplementation. | at 0h, 72h, day7, day 14, every other week until postmenstrual age 29 week and thereafter 30, 32, 34, 36 and 40 weeks postmenstrual age
  Postnatal serum fatty acid composition
Postnatal brain development, as assessed by Magnetic Resonance Imaging (MRI) | at 40 weeks postmenstrual age and at 2.0 y corrected age and 5.5 y uncorrected age.
  Postnatal brain development, as assessed by Magnetic Resonance Imaging (MRI), Volumetric and Diffusor Tensor Imaging (DTI).
Outcome in p-glucose | at 0h, 72h, day7, day 14, every other week until postmenstrual age 29 week and thereafter at 30, 32, 34, 36 and 40 weeks postmenstrual age.
  Neonatal glucose metabolism.
Outcome in weight in kilograms. | at day 0, 7, 14, 21 and thereafter every week up to 40 weeks postmenstrual age
  Postnatal growth development, weight in kilograms.
Outcome in head circumference in centimeters. | at day 0, 7, 14, 21 and thereafter every week up to 40 weeks postmenstrual age
  Postnatal growth development, head circumference in centimeters.
Outcome in height in centimeters. | at day 0, 7, 14, 21 and thereafter every week up to 40 weeks postmenstrual age
  Postnatal growth development, height in centimeter.
Outcome of neonatal morbidities. | Reported as adverse event from birth to 40 weeks postmenstrual age.
  Frequency of neonatal morbidities such as bronchopulmonary dysplasia (BPD), cerebral intraventricular hemorrhage (IVH), patent ductus arteriosus (PDA), sepsis and necrotizing enterocolitis (NEC).

CONTACTS AND LOCATIONS:
Overall Officials: Ann ca Hellstrom, Professor, Principal Investigator — Göteborg University; David Ley, Professor, Principal Investigator — University of Lund; Boubou Hallberg, MD,PhD, Principal Investigator — University of Karolinska; Karin Savman, MD, PhD, Principal Investigator — Göteborg University
Locations (3):
- Sweden (3):
  - Queen Silvias Childrens Hospital, Gothenburg
  - Skanes Universitetssjukhus, Lund
  - KI, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hellstrom W, Lundgren P, Nilsson AK, Nilsson S, Hard AL, Sjobom U, Lofqvist C, Bjorkman-Burtscher IM, Wackernagel D, Hansen-Pupp I, Smith LE, Hallberg B, Savman K, Ley D, Hellstrom A, Heckemann RA. Effect of enteral arachidonic acid and docosahexaenoic acid supplementation on brain volumes at term in preterm infants: a secondary outcome analysis of a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2026 Jan 19:fetalneonatal-2024-328292. doi: 10.1136/archdischild-2024-328292. Online ahead of print. PMID 41554627
- [Derived] Lundgren P, Danielsson H, Panwar MB, Alvez MB, Pivodic A, Zhong W, Brusselaers N, Wackernagel D, Sjobom U, Savman K, Pupp IH, Ley D, Klevebro S, Nilsson AK, Fu Z, Smith LEH, Uhlen M, Hellstrom A. Proteomic Profile in Retinopathy of Prematurity: A Secondary Analysis of the Mega Donna Mega Randomized Clinical Trial. JAMA Ophthalmol. 2026 Jan 8:e255594. doi: 10.1001/jamaophthalmol.2025.5594. Online ahead of print. PMID 41505112
- [Derived] Klevebro S, Kebede Merid S, Sjobom U, Zhong W, Danielsson H, Wackernagel D, Hansen-Pupp I, Ley D, Savman K, Uhlen M, Smith LEH, Hellstrom A, Nilsson AK. Arachidonic acid and docosahexaenoic acid levels correlate with the inflammation proteome in extremely preterm infants. Clin Nutr. 2024 May;43(5):1162-1170. doi: 10.1016/j.clnu.2024.03.031. Epub 2024 Apr 3. PMID 38603973
- [Derived] Sjobom U, Andersson MX, Pivodic A, Lund AM, Vanpee M, Hansen-Pupp I, Ley D, Wackernagel D, Savman K, Smith LEH, Lofqvist C, Hellstrom A, Nilsson AK. Modification of serum fatty acids in preterm infants by parenteral lipids and enteral docosahexaenoic acid/arachidonic acid: A secondary analysis of the Mega Donna Mega trial. Clin Nutr. 2023 Jun;42(6):962-971. doi: 10.1016/j.clnu.2023.04.020. Epub 2023 Apr 17. PMID 37120902
- [Derived] Pivodic A, Johansson H, Smith LE, Lofqvist C, Albertsson-Wikland K, Nilsson S, Hellstrom A. Evaluation of the Retinopathy of Prematurity Activity Scale (ROP-ActS) in a randomised controlled trial aiming for prevention of severe ROP: a substudy of the Mega Donna Mega trial. BMJ Open Ophthalmol. 2022 Apr 8;7(1):e000923. doi: 10.1136/bmjophth-2021-000923. eCollection 2022. PMID 35495419
- [Derived] Hortensius LM, Hellstrom W, Savman K, Heckemann RA, Bjorkman-Burtscher IM, Groenendaal F, Andersson MX, Nilsson AK, Tataranno ML, van Elburg RM, Hellstrom A, Benders MJNL. Serum docosahexaenoic acid levels are associated with brain volumes in extremely preterm born infants. Pediatr Res. 2021 Dec;90(6):1177-1185. doi: 10.1038/s41390-021-01645-w. Epub 2021 Aug 14. PMID 34392310
- [Derived] Hellstrom A, Nilsson AK, Wackernagel D, Pivodic A, Vanpee M, Sjobom U, Hellgren G, Hallberg B, Domellof M, Klevebro S, Hellstrom W, Andersson M, Lund AM, Lofqvist C, Elfvin A, Savman K, Hansen-Pupp I, Hard AL, Smith LEH, Ley D. Effect of Enteral Lipid Supplement on Severe Retinopathy of Prematurity: A Randomized Clinical Trial. JAMA Pediatr. 2021 Apr 1;175(4):359-367. doi: 10.1001/jamapediatrics.2020.5653. PMID 33523106